CLINICAL TRIAL: NCT00716404
Title: Post-Market Observational Study of Intra-Renal Drug Delivery
Acronym: PROVIDE
Status: Withdrawn | Type: Observational
Why Stopped: FlowMedica was purchased by AngioDynamics. Study will be re-started by AngioDynamics.
Sponsor: FlowMedica, Inc. (Industry)
Responsible Party: Burt Goodson/Director, Scientific Affairs, AngioDynamics, Inc.
Other Study IDs: CL0015
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Targeted Renal Therapy
Keywords: FlowMedica; Benephit; TRT; Patients; Components; Benephit Infusion System; Planned; To be used

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All (consecutive) patients in whom one or more components of the Benephit Infusion System are planned to be used are eligible for enrollment in the study and should be offered informed consent.
  Interventions: Device: Targeted Renal Therapy

INTERVENTIONS:
Device: Targeted Renal Therapy — Patient diagnosis, treatment, and follow-up are left to the discretion of the participating investigator. There are no requisites as to how patients should be managed as this is intended to be an observational study. No procedures other than usage of the Benephit Infusion System per its Instructions for Use are specifically required for participation in this study.
  Other Names: Benephit CV Infusion System; Benephit PV Infusion System; Benephit PVMini Infusion System; Benephit PVSolo Infusion System; Benephit XT Infusion System

SUMMARY:
This is a prospective, observational, multi-center study with consecutive enrollment. Up to 1,000 patients will be enrolled. The objective of this post-marketing surveillance study is to collect clinical usage patterns of the Benephit Infusion Systems. As a result, FlowMedica will be able to:

1. Better understand and quantify usage patterns including patient characteristics, adjunctive procedures, and infusion agents.
2. Collect user-interface information and overall customer satisfaction.
3. Monitor post-marketing device performance.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to one or more components of the Benephit Infusion System
* Ability to give written informed consent

Exclusion Criteria:

* Inclusion in another clinical study that may affect usage of the Benephit system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients in whom one or more components of the Benephit Infusion System are planned to be used.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: James A Tumlin, MD, Principal Investigator — Southeast Renal Associates; David E Allie, MD, Principal Investigator — Cardiovascular Institute of the South
Locations (4):
- United States (4):
  - Scripps Clinic, La Jolla, California
  - Owensboro Heart & Vascular, Owensboro, Kentucky
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Providence Heart & Vascular, Portland, Oregon

REFERENCES:
- See also: Sponsor Website — http://www.flowmedica.com